CLINICAL TRIAL: NCT05974631
Title: A Hybrid Effectiveness-Implementation Trial of Treatments for Veterans With PTSD at Elevated Acute Risk for Suicide
Brief Title: Evaluating Treatments for Suicidal Veterans With PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDR 22-185
Record Dates: First submitted 2023-07-05; First posted 2023-08-03 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Self-directed Violence; Post-traumatic Stress Disorder (PTSD)
Keywords: Stress Disorders, Post-Traumatic; Suicide; Self-Injurious Behavior
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicide; Self-Injurious Behavior | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Intervention Model Description: 2-arm randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be masked to participants' treatment condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DBT + DBT PE (Experimental): This condition combines one year of standard Dialectical Behavior Therapy (DBT) with the DBT Prolonged Exposure (DBT PE) protocol for PTSD.
  Interventions: Behavioral: Dialectical Behavior Therapy; Behavioral: Dialectical Behavior Therapy Prolonged Exposure protocol
- PE + SRM (Active Comparator): This condition provides up to 18 sessions of Prolonged Exposure therapy (PE) for PTSD augmented with suicide risk management (SRM).
  Interventions: Behavioral: Prolonged Exposure therapy; Behavioral: Suicide risk management

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy — Standard Dialectical Behavior Therapy (DBT), including DBT individual therapy (1 hour/week), DBT group skills training (2 hours/week), between-session coaching (as needed during business hours), and therapist consultation team (1-1.5 hours/week).
  Other Names: DBT
  Arms: DBT + DBT PE
Behavioral: Dialectical Behavior Therapy Prolonged Exposure protocol — DBT PE is designed to be integrated into DBT to formally treat PTSD once patients meet standardized readiness criteria. The core procedures are in vivo and imaginal exposure with processing that are delivered in individual therapy sessions (1.5 hours/week).
  Other Names: DBT PE
  Arms: DBT + DBT PE
Behavioral: Prolonged Exposure therapy — Standard PE is delivered in individual therapy sessions (1.5 hours/week) and uses the core procedures of in vivo and imaginal exposure with processing.
  Other Names: PE
  Arms: PE + SRM
Behavioral: Suicide risk management — Standard VA suicide risk management procedures, including comprehensive suicide risk assessment and safety planning.
  Other Names: SRM
  Arms: PE + SRM

SUMMARY:
Posttraumatic Stress Disorder (PTSD) is a significant driver of suicide risk among Veterans, but there is a critical knowledge gap about how to treat PTSD among people at elevated risk for suicide. Although evidence-based treatments for PTSD reduce suicide risk, Veterans at high risk for suicidal behavior rarely receive these potentially life-saving treatments. Prior research suggests that a treatment that combines Dialectical Behavior Therapy (DBT) with the DBT Prolonged Exposure protocol (DBT PE) for PTSD improves both PTSD and suicide-related outcomes. This study will evaluate whether DBT + DBT PE improves these outcomes more than Prolonged Exposure plus suicide risk management, the gold standard VA care for this population. The proposed study will also examine factors that make it easier and harder to implement these treatments in VA settings. The results will help to inform treatment guidelines for this high-priority Veteran population.

DETAILED DESCRIPTION:
Background: Posttraumatic stress disorder (PTSD) is a significant risk factor for suicide among Veterans. Evidence-based psychotherapies (EBPs) for PTSD reduce suicide risk, but Veterans at elevated acute risk for suicide, such as those who have engaged in self-directed violence (SDV), rarely receive these treatments. This is largely due to the historical exclusion of high-risk individuals from PTSD treatment trials, which has resulted in a lack of evidence-based guidance about indicated treatments for this population. Without such guidance, clinicians are often reluctant to use EBPs for PTSD with suicidal individuals. A treatment that combines Dialectical Behavior Therapy (DBT), a suicide-focused EBP, with the DBT Prolonged Exposure (DBT PE) protocol for PTSD has been developed for this high-risk population and shows promise in reducing both SDV and PTSD while being feasible, acceptable, and safe to deliver. However, a large-scale randomized controlled trial (RCT) is needed. This study will compare the effectiveness of DBT + DBT PE to the current VHA gold standard of care for this population, Prolonged Exposure therapy augmented with suicide risk management (PE + SRM), while also examining the potential for implementation of both interventions in VHA.

Significance: There is a critical gap in knowledge about how to treat PTSD among individuals at high risk for suicidal behavior. As a result, VA/DoD Clinical Practice Guidelines do not specify indicated treatment strategies for this population. Experts have recommended two approaches to facilitate the safe and effective use of EBPs for PTSD with individuals at elevated acute suicide risk, including combining these treatments with suicide-focused EBPs or augmenting them with suicide risk management strategies. This project will help to fill this critical gap by rigorously evaluating these two approaches among Veterans with SDV. The results will provide important information to inform guidelines about indicated treatments for this high-risk population.

Innovativeness: This will be the first large-scale RCT to evaluate treatments for PTSD among Veterans who have engaged in SDV, an HSR&D high priority group. The DBT + DBT PE intervention is the first treatment designed to address both SDV and PTSD, and results will indicate if this novel treatment improves outcomes compared to the current VHA gold standard of care. To facilitate more rapid implementation of these findings into clinical practice, implementation barriers and facilitators for both treatments will also be evaluated.

Specific Aims: This study will randomize 125 Veterans with PTSD, recent and repeated SDV, current suicidal ideation, and emotion dysregulation to DBT + DBT PE (intervention) or PE + SRM (control). Aim 1 will test the hypothesis that DBT + DBT PE will be superior to PE + SRM in improving clinical outcomes and engagement in trauma-focused treatment. Exploratory analyses will examine Veteran characteristics that may predict better engagement and outcomes in DBT + DBT PE versus PE + SRM. Aim 2 will examine barriers and facilitators to implementation of both treatments.

Methods: This is a multi-site hybrid type 1 effectiveness-implementation trial. Veterans will be treated in outpatient settings at three VA sites and assessed at 5 points over 16 months. A mixed-methods approach will be used to evaluate barriers and facilitators to implementation, including conducting interviews with 45 key stakeholders (Veterans, providers, and leadership).

Primary Outcomes/Endpoints: Primary outcomes will be reductions in SDV episodes at 16-month follow-up and reductions in PTSD severity at post-treatment.

Implementation/Next Steps: This project will provide much-needed information about how to safely and effectively treat PTSD among Veterans at elevated acute risk for suicide. If one or both treatments are found effective, Aim 2 will provide vital information about how to maximize future implementation success. Future implementation activities would be coordinated with the investigators' national operational partners.

ELIGIBILITY:
Inclusion Criteria:

* PTSD
* Recent and repeated self-directed violence
* Current suicidal ideation
* Emotion dysregulation
* Veteran eligible for VHA mental health care at participating site
* Age 18+
* Willing to participate in all study activities

Exclusion Criteria:

* Unable to maintain safety independently
* Currently engaged in and/or recent (past year) history of receiving a sufficient dose of DBT or PE
* Plan to move away or be unavailable for >4 weeks in the next 18 months
* Unable to sufficiently comprehend study procedures due to lack of English proficiency or moderate to severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Self-Injurious Thoughts and Behaviors Interview - Revised Short Form (SITBI-R-SF) | Baseline to 16 months
  Number of self-directed violence episodes
Clinician-Administered PTSD Scale for DSM-5 Revised (CAPS-5-R) | Baseline to 16 months
  Total Severity Score (range = 0 - 200, higher is worse)

SECONDARY OUTCOMES:
Columbia - Suicide Severity Rating Scale (C-SSRS), Suicide Ideation subscales | Baseline to 16 months
  Total Score (range = 0 - 5, higher is worse)
PROMIS Global Mental Health | Baseline to 16 months
  Total Score (range = 4 - 20, higher is better)
Difficulties in Emotion Regulation Scale-16 (DERS-16) | Baseline to 16 months
  Total Score (range = 16 - 80, higher is worse)
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Baseline to 16 months
  General Disability Score (range = 12 - 60, higher is worse)
Self-Injurious Thoughts and Behaviors Interview Revised Short Form (SITBI-R-SF) | Baseline to 16 months
  Non-suicidal self-injury frequency and remission; Suicide attempt frequency and remission
Clinician-Administered PTSD Scale for DSM-5 Revised (CAPS-5-R) | Baseline to 16 months
  PTSD diagnostic status

OTHER OUTCOMES:
Treatment History Interview (THI) | Baseline to 16 months
  Non-VA psychotherapy, psychiatric crisis services, and psychotropic medications
VA Service Use Form | Baseline to 16 months
  VA mental health service use and psychotropic medications
Credibility Expectancy Questionnaire (CEQ) | Baseline to 16 months
  Total score (range = 1 - 7, higher is better)
Client Satisfaction Questionnaire (CSQ) | Post-treatment (4 months in PE + SRM, 12 months in DBT + DBT PE)
  Total score (range = 8 - 32, higher is better)
Dissociative Experiences Scale - Taxon (DES-T) | Baseline to 16 months
  Total score (range = 0 - 80, higher is worse)
Trauma-Related Shame Inventory (TRSI) | Baseline to 16 months
  Total score (range = 0 - 72, higher is worse)
Self-Compassion Scale (SCS) | Baseline to 16 months
  Total score (range = 1 - 5, higher is better)
Borderline Symptom List - Behavioral Supplement (BSL-BS) | Baseline to 16 months
  Total score (range = 0 - 44, higher is worse)
PTSD Checklist for DSM-5 (PCL-5) | Baseline to 16 months
  Total severity score (range = 0 - 80, higher is worse)
Post-Traumatic Cognitions Inventory-9 (PTCI-9) | Baseline to 16 months
  Total score (range = 9 to 63, higher is worse)
PROMIS Sadness | Baseline to 16 months
  Total score (range = 8 - 40, higher is worse)
PROMIS Fear-Affect | Baseline to 16 months
  Total score (range = 7 - 35, higher is worse)
PROMIS Anger-Affect | Baseline to 16 months
  Total score (range = 5 - 25, higher is worse)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie S Harned, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (4):
- United States (4):
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified, anonymized data that underlie results in a publication may be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Starting after publication of relevant data
Access Criteria: Data may be shared in response to written requests submitted to the PI by other researchers. Such data sharing will take place under a written agreement that prohibits the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are in the dataset.